CLINICAL TRIAL: NCT06789861
Title: A First in Human, Three-part, Double Blind, Randomized, Placebo-controlled, Single and Multiple Ascending Dose Study to Investigate Safety and Pharmacokinetics of TT5 in Healthy Participants and Surgical Patients
Brief Title: A First in Human Study of TT5 in Single and Multiple Ascending Doses in Healthy Volunteers and Surgical Patients
Acronym: TAFA-FIRST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tafalgie Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-TT5-PH1-001
Record Dates: First submitted 2025-01-09; First posted 2025-01-23 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TT5 (Experimental)
  Interventions: Drug: TT5
- TT5 vehicle (Placebo Comparator)
  Interventions: Drug: Placebo - TT5 vehicle

INTERVENTIONS:
Drug: TT5 — Direct Intravenous administration of TT5 (5 ascending doses in Single Ascending Dose Part and 3 ascending doses administered during 7 days in Multiple Ascending Dose Part in healthy volunteers) Direct Intravenous administration of TT5 in surgical patients (4 doses administered on the same day) in surgical patients
  Arms: TT5
Drug: Placebo - TT5 vehicle — Intravenous administration of vehicule, according to the same drug regimen than TT5
  Arms: TT5 vehicle

SUMMARY:
This study is a First in Human, three-parts, double-blind, randomized, placebo-controlled, single and multiple ascending dose study. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of TT5 at different doses in healthy and surgical participants.

DETAILED DESCRIPTION:
The study will be divided into three parts:

Part A: Single Ascending Dose - healthy participants cohorts with up to 5 dose levels.

Part B: Multiple Ascending Doses - healthy participants cohorts with up to 3 dose levels.

Part C: Surgical patients cohorts with up to 3 dose levels.

The primary Objective is to investigate the safety and tolerability of TT5 in single and multiple ascending intravenous doses in healthy participants and in surgical patients.

The Secondary Objectives are To investigate the pharmacokinetics (PK) of TT5 after single and multiple ascending intravenous doses in healthy participants and after intravenous doses in surgical patients.

* To investigate the acute and chronic psychological subjective response of the healthy participants and surgical patients to TT5
* To assess the pharmacodynamics (PD) of TT5 after intravenous doses in surgical patients. Exploratory Objectives areto explore potential fluid biomarkers for TT5

ELIGIBILITY:
Main inclusion criteria for Parts A and B:

* Non-smoker for the confinement period of the study.
* Medically healthy and without clinically significant abnormalities.
* Negative screen for alcohol and drugs of abuse.
* No history of psychiatric disorders.
* Female participants of non-childbearing potential must be post-menopausal or surgically sterile at least 3 months prior to dosing.
* Sexually active females of childbearing potential and non-sterile males must be willing to use an acceptable contraceptive method throughout the study.
* Able to understand the study procedures and provide signed informed consent to participate in the study in English.

Main exclusion criteria for Parts A and B:

* History of clinically significant asthma, anaphylaxis, major medical, psychiatric illness or surgery.
* Acute or chronic clinically relevant systemic disease or disorder.
* Renal insufficiency
* History of drug or alcohol consumption abuse.
* Drinking excessive amounts of tea, coffee, chocolate and/or beverage containing caffeine.
* Have used any investigational drug or participated in any clinical trial within 4 weeks prior to screening.
* Unable to refrain from strenuous exercise.
* Participant who has received blood or plasma derivatives, who had a surgery or who has given blood within 4 weeks prior to the screening visit or has planned to give blood or sperm within the 90 days following the study.
* Pregnant or lactating female participant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and serious adverse events (SAEs) | SAD cohorts: Day-1 through Day 8; MAD cohorts: Day-1 through Day 14
  Number of AEs and SAEs:To investigate the safety and tolerability of TT5
Clinically significant changes in physical examinations | SAD cohorts: Baseline through Day 8; MAD cohorts: Baseline through Day 14
  % of participants with clinically significant changes from baseline in physical examinations by measuring general appearance, head, eyes, ears, nose, throat (HEENT), neck (including thyroid and nodes), cardiovascular, respiratory, gastrointestinal, renal, neurological, musculoskeletal, and skin.
Clinically significant changes in vital signs | SAD cohorts: Day-1 through Day 8; MAD cohorts: Day-1 through Day 14
  % of participants with clinically significant change from baseline in vital signs by measuring heart rate, blood pressure, temperature, and respiratory rate
Clinically significant changes in laboratory analysis | SAD cohorts: Day-1 through Day 8; MAD cohorts: Day-1 through Day 14
  Mean and SD of clinically significant changes from baseline in laboratory analysis including hematology, coagulation, biochemistry, and urinalysis
Bond and Lader Visual Analog Scale (VAS) | SAD cohorts: Day 1 through Day 8; MAD cohorts: Day 1 through Day 14
  VAS item values: To assess vigilance will using a Visual Analogic Scale namely the Bond-Lader VAS of Mood and Alertness

SECONDARY OUTCOMES:
Plasma AUC0-t measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Area under the concentration-time curve from time zero until the last observed concentration (AUC0-t) h*ng/ml
Plasma AUC0-inf measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Area under the concentration-time curve from time zero to infinity (AUC0-inf) h*ng/ml
Plasma Cmax measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Maximum concentration measurement in plasma (ng/ml)
Plasma Tmax measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Time to maximum observed concentration in plasma (hours)
Plasma T½ el measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Terminal elimination half-life (T½ el) in plasma (hours)
Plasma Kel measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Terminal elimination rate constant (Kel) in plasma (fraction/h)
Plasma Cl/F measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Apparent clearance (Cl/F) in plasma (mL/min)
Plasma Vz/F measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Apparent volume of distribution (Vz/F) in plasma (liters)
Urine CLr measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Renal clearance measurement in urine (mL/min)
Urine Aet1-t2 measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Amount excreted in urine (Aet1-t2) per interval (mL/min)
Urine Ae0-t measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Cumulative urinary excretion from time zero to time t (Ae0-t) ( (mL/min)
Urine Ae%dose measurement | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  % of drug recovered in urine (Ae%dose)
ARCI | SAD cohorts: Day 1 through Day 8; MAD cohorts: Day 1 through Day 14
  Total Score and Sub-scores of Addiction Research Center Inventory questionnaire to investigate subjective effects

OTHER OUTCOMES:
Biomarkers | SAD cohorts: Day 1 through Day 2; MAD cohorts: Day 1 through Day 8
  Fluid Biomarkers concentration (pmol/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Ludbrook, MD, Principal Investigator — University of Adelaide and Royal Adelaide Hospital.
Locations (1):
- Cmax & PARC, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No